CLINICAL TRIAL: NCT00559741
Title: Phase 2 Study to Improve Tolerance of Chemotherapy Involving Cetuximab and Multidrug FOLFIRI, With Pharmacokinetic and Pharmacogenetic Studies, in Patients With Metastatic Colorectal Cancer
Brief Title: Cetuximab and Combination Chemotherapy in Treating Patients With Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574065; CPP-FOLFIRICETUX; INCA-RECF0108
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; recurrent colon cancer; stage IV rectal cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Biological: cetuximab
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Other: pharmacological study

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as irinotecan, fluorouracil, and leucovorin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cetuximab together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with combination chemotherapy works in treating patients with advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Improve hematologic and gastrointestinal tolerance to cetuximab and irinotecan hydrochloride, fluorouracil, and leucovorin calcium (FOLFIRI) in patients with advanced or metastatic colorectal cancer.

Secondary

* Increase the effectiveness of this regimen by intensifying the treatment.
* Specify the constitutional genetic and genomic tumor parameters that could interfere with and predict the toxicity and/or antitumor efficacy of this regimen.
* Assess the time to progression.

OUTLINE: This is a multicenter study.

Patients receive irinotecan hydrochloride IV over 90 minutes, leucovorin calcium IV over 2 hours, and cetuximab IV over 1-2 hours on day 1. Patients also receive fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

Pharmacokinetic and pharmacogenetic studies are also conducted.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Advanced or metastatic disease
* Scheduled to receive first- or second-line therapy for metastatic disease
* No cerebral metastases or symptomatic or uncontrolled meningeal disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Alkaline phosphatase ≤ 5 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No intestinal blockage
* No complete dihydropyrimidine dehydrogenase deficiency
* No chronic inflammatory disease of the colon
* No other cancer except for nonmelanoma skin cancer or curatively treated carcinoma of the cervix or breast
* No other severe condition, or condition that is likely to worsen, including any of the following:

  * Unstable heart disease
  * Myocardial infarction within the past 6 months
  * Active uncontrolled infection
* No contraindication to atropine

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior anticancer therapy
* More than 4 weeks since prior and no other concurrent investigational therapy
* Prior adjuvant chemotherapy allowed
* No prior fluorouracil or irinotecan hydrochloride
* No other concurrent anticancer therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-10; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Improvement of hematologic and gastrointestinal tolerance to therapy

SECONDARY OUTCOMES:
Efficacy
Genetic and genomic tumor parameters that could interfere with and predict the toxicity and/or antitumor efficacy of therapy
Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Erick Gamelin, MD, Study Chair — Institut Cancerologie de l'Ouest
Locations (1):
- Centre Paul Papin, Angers, France

REFERENCES:
- [Result] Rouits E, Charasson V, Petain A, Boisdron-Celle M, Delord JP, Fonck M, Laurand A, Poirier AL, Morel A, Chatelut E, Robert J, Gamelin E. Pharmacokinetic and pharmacogenetic determinants of the activity and toxicity of irinotecan in metastatic colorectal cancer patients. Br J Cancer. 2008 Oct 21;99(8):1239-45. doi: 10.1038/sj.bjc.6604673. Epub 2008 Sep 16. PMID 18797458
- [Derived] Lobet S, Paintaud G, Azzopardi N, Passot C, Caulet M, Chautard R, Desvignes C, Capitain O, Tougeron D, Lecomte T, Ternant D. Relationship Between Cetuximab Target-Mediated Pharmacokinetics and Progression-Free Survival in Metastatic Colorectal Cancer Patients. Clin Pharmacokinet. 2023 Sep;62(9):1263-1274. doi: 10.1007/s40262-023-01270-2. Epub 2023 Jul 13. PMID 37442917
- [Derived] Rollin J, Payance A, Gouilleux-Gruart V, Boisdron-Celle M, Azzopardi N, Morel A, Gruel Y, Paintaud G, Gamelin E, Watier H, Lecomte T. Significant effect of VEGFA polymorphisms on the clinical outcome of metastatic colorectal cancer patients treated with FOLFIRI-cetuximab. Pharmacogenomics. 2015 Dec;16(18):2035-43. doi: 10.2217/pgs.15.139. Epub 2015 Nov 30. PMID 26615857